CLINICAL TRIAL: NCT06760780
Title: Effect of Scenario-based Teaching on Osteoporosis Awareness in Nursing Students: a Randomized Controlled Trial
Brief Title: Osteoporosis Awareness Among Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cavusoglu, Doctorate, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MersinUni.
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Interventional
Keywords: Scenario-supported education; Nursing students; Osteoporosis awareness

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since the nursing students participating in the study will be in either the experimental or control group, they will not be blinded, and the researchers will only be blinded during group assignment. The data will be entered into the computer by the researchers and a biostatistician independent of the study will analyze the data and report the results without knowing which groups are experimental or control. The biostatistician will therefore be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: Scenario group (Experimental): Theoretical lesson on osteoporosis and a scenario example on osteoporosis will be covered with the experimental group.
  Interventions: Other: Experimental
- Other: Control group (Other): The control group will be given a theoretical lesson on osteoporosis. No additional intervention will be made.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The experimental group will first be given a theoretical lesson prepared in line with the current literature on osteoporosis. At the end of the lesson, a prepared scenario example on osteoporosis will be covered.
  Arms: Experimental group: Scenario group
Other: Control — The control group will only be given a theoretical lesson prepared in line with the current literature on osteoporosis. No other intervention will be made.
  Arms: Other: Control group

SUMMARY:
The aim of this clinical study is to determine the effect of scenario-based training of nursing students on awareness of osteoporosis.

To this end, the most important questions to be answered in the study are

* What is the level of osteoporosis awareness among nursing students at the start of the study?
* Does scenario-based education have an impact on osteoporosis awareness?

Participants:

All student nurses participating in the study will first receive theoretical training on osteoporosis. At the end of the training, a scenario example prepared by the researchers on the topic of osteoporosis is worked on with the students in the experimental group. No additional intervention is carried out with the control group.

DETAILED DESCRIPTION:
In this study, 78 nursing students randomly assigned to the experimental and control groups are first interviewed using the personal information questionnaire and the Osteoporosis Awareness Scale. This is followed by a four-hour theoretical lesson prepared by the researchers in accordance with current literature and textbooks on osteoporosis as part of the Joint and Connective Tissue Diseases and Nursing course. At the end of the theoretical lessons, a scenario example prepared by the researchers, again using current literature and case presentations, will be worked on with the students in the experimental group. No other application is made for the control group. The Personal Information Questionnaire and the Osteoporosis Awareness Scale will be re-administered to both groups four weeks after the end of the theoretical lesson.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above,
* Mersin University Faculty of Nursing 2nd year students,
* Have not received any other training on osteoporosis before,
* Willing to participate in the research,
* Have cognitive competence to fill out the data collection form,
* Those who sign the Informed Voluntary Consent Form will be included.

Exclusion Criteria:

* Those under the age of 18,
* Not a 2nd year student at Mersin University Faculty of Nursing,
* Have previously received different training on osteoporosis,
* Do not want to participate in the research,
* Do not have the cognitive ability to fill out the data collection form,
* Those who do not sign the Informed Consent Form will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis awareness level will be assessed using the Osteoporosis Awareness Scale. | Change from before implementation and 4th week of practice
  The Osteoporosis Awareness Scale consists of 31 items and 5 subscales. Responses to scale items are rated on a 4-point Likert-type scale ranging from 1 to 4 (4 = I know very well, 3 = I know, 2 = I know a little, 1 = I don't know at all). The lowest and highest possible scores from the scale are 31 and 124, respectively. The higher the average score obtained from the overall scale, the higher the osteoporosis awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Çavuşoğlu, Doctorate, Study Director — Mersin University; Meral Gün, Doctorate, Principal Investigator — Mersin University

IPD SHARING:
Plan to Share IPD: No